CLINICAL TRIAL: NCT02245438
Title: A Single Centre, Open-label, Randomized, Parallel Group, Multiple Dose Comparison of the Effect of TPV 750 mg and RTV 200 mg or TPV 500 mg and RTV 100 mg, Administered Twice Daily, on the Pharmacokinetic Characteristics of Norethindrone-Ethinyl Estradiol (Ortho®-1/35 ) Administered as a Single Dose, in Healthy Female Adult Volunteers.
Brief Title: Effect of Tipranavir and Ritonavir on the Pharmacokinetic Characteristics of Norethindrone-Ethinyl Estradiol in Healthy Female Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.22
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; ovcon 35

ARMS (2):
- TPV/RTV low dose (Experimental)
  Interventions: Drug: Tipranavir low dose; Drug: Ritonavir low dose; Drug: Norethindrone-Ethinyl Estradiol
- TPV/RTV high dose (Experimental)
  Interventions: Drug: Tipranavir high dose; Drug: Ritonavir high dose; Drug: Norethindrone-Ethinyl Estradiol

INTERVENTIONS:
Drug: Tipranavir low dose
  Arms: TPV/RTV low dose
Drug: Tipranavir high dose
  Arms: TPV/RTV high dose
Drug: Ritonavir low dose
  Other Names: Norvir-SEC®
  Arms: TPV/RTV low dose
Drug: Ritonavir high dose
  Other Names: Norvir-SEC®
  Arms: TPV/RTV high dose
Drug: Norethindrone-Ethinyl Estradiol
  Other Names: Ortho®-1/35

SUMMARY:
Study to characterize the effects of two dose combinations of Tipranavir (TPV)/Ritonavir (RTV) (TPV 750 mg/RTV 200 mg and TPV 500 mg/RTV 100 mg), administered twice-daily, on the pharmacokinetics of Norethindrone-Ethinyl Estradiol (NET/EE) 1 mg/ 0.035 mg administered as a single dose.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects between 18 and 50 years of age inclusive
2. A Body Mass Index (BMI) between 18 and 29 kg/m2
3. Signed informed consent prior to trial participation
4. Ability to swallow numerous large capsules without difficulty
5. Acceptable laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity is less than or equal to Grade 1, based on the AIDS Clinical Trials Group Grading Scale. All abnormal laboratory values greater than Grade 1 are subject to approval by the trial clinical monitor.
6. Acceptable medical history, physical examination and ECG, and chest X-ray (if not conducted within the last 12 months) are required prior to entering the treatment phase of the study
7. Willingness to abstain from alcohol for 48 hours prior to Study Day 0 and abstain from alcohol for the duration of the study. In addition, red wine must not have been ingested within 5 days prior to Day 0 (Visit 2)
8. Willingness to abstain from ingesting grapefruit, grapefruit juice, or products containing grapefruit juice, within 10 days before Day 0, Visit 2 and for the duration of the study
9. Willingness to abstain from ingesting Seville oranges, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc) within 5 days of Day 0, Visit 2 and for the duration of the study
10. Willingness to abstain from over the counter herbal medications for the duration of the study
11. Reasonable probability for completion of the study

Exclusion Criteria:

1. Female subjects who are of reproductive potential who:

   * Have positive serum beta-human chorionic gonadotropin at Visit 1, or on Day 0 or Day 1
   * Have not been using a barrier contraceptive method for at least 3 months prior to Visit 3 (Day 1)
   * Are not willing to use a reliable method of double-barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during the trial and 30 days after completion/termination
   * Are breast-feeding
2. Participation in another trial with an investigational medicine within 30 days prior to Day 0 (Visit 2)
3. Use of any medication listed in the protocol within 30 days prior to Day 0 (Visit 2)
4. Use of any other pharmacological contraceptive (including oral, patch or injectable contraceptives) for 1 month prior to study initiation and for the duration of the study
5. Administration of antibiotics within 10 days prior to Day 0 (Visit 2) or during the trial
6. History of central nervous system (CNS), gastrointestinal, hepatic, or renal disorders within the past sixty (60) days. Subjects will be excluded for these disorders greater than sixty days if, in the opinion of the investigator, the subject does not qualify as a healthy volunteer
7. History of thrombotic disease
8. History of migraine headache
9. Have serological evidence of hepatitis B or C virus
10. Have serological evidence of exposure to HIV
11. Recent history of alcohol or substance abuse (within 6 months of study period)
12. Cigarette smoking (greater than 10 cigarettes per day)
13. Blood or plasma donations within 30 days prior to Day 0 (Visit 2) or during the trial.
14. Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min. For subjects with a resting heart rate below 50, due to a high fitness level, the investigator may discuss exclusion with the medical monitor on a case-by-case basis
15. Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering Tipranavir, Ritonavir or NET/EE to the subject
16. Subjects who have had an acute illness within 2 weeks prior to Day 0 (Visit 2)
17. Subjects who are currently taking any over-the-counter drug within 7 days prior to Day 0,(Visit 2) or who are currently taking any prescription drug that, in the opinion of the investigator in consultation with the clinical monitor, might interfere with either the absorption, distribution or metabolism of the test substances
18. Known hypersensitivity to TPV, RTV, or NET/EE
19. Inability to comply with the protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2002-05; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve | up to day 17
Maximum plasma concentration of the analyte | up to day 17
Drug concentration of the analyte in plasma at 12 hours after administration | up to day 17

SECONDARY OUTCOMES:
Oral clearance of the analyte | up to day 17
Time of maximum concentration of the analyte | up to day 17
Apparent terminal half life of the analyte | up to day 17
Number of subjects with adverse events | up to 45 days
Number of subject with clinically relevant changes in laboratory parameters | up to 17 days